CLINICAL TRIAL: NCT03804827
Title: Impact of Sleep Disordered Breathing on Cardiac Injury in Acutely Decompensated Congestive Heart Failure
Brief Title: Sleep Disordered Breathing in Acute Congestive Heart Failure
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Assistant Professor, University of California, San Diego
Other Study IDs: 181121
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Obstructive Sleep Apnea; Heart Failure; With Decompensation
Keywords: Sleep; OSA; CSA; CHF; Heart Failure; Troponin
MeSH Terms: conditions — Sleep Apnea, Obstructive; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum retention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Failure With Sleep Disordered Breathing: AHI3% >/= 5 events per hour of sleep.
- Heart Failure without Sleep Disordered Breathing: AHI3% < 5 events per hour of sleep.

SUMMARY:
The goal of this study is to determine if sleep disordered breathing results in a measurable degree of overnight myocardial stress/injury in patients with acutely decompensated congestive heart failure. A secondary goal is to determine of a period of medical management attenuates this sleep disordered breathing-induced cardiac injury in this patient population.

DETAILED DESCRIPTION:
Consecutive patients admitted to the hospital with acutely decompensated heart failure will be identified for potential enrollment in this study. Enrolled patients will first be asked to complete questionnaires to assess their symptoms and risk of having sleep apnea.

Relevant information will be obtained from the electronic medical record (age, gender, body mass index, co-morbidities, medications, prior echocardiography results). Subjects will then undergo a "type III" portable monitoring sleep study on the first or second night of their hospital admission, which measures respiratory effort, nasal airflow, oxyhemoglobin saturation, and heart rate. Blood samples will be collected on the evening before (08:00 PM +/- 2 hours), and the morning after (06:00 AM +/-2 hours) sleep apnea testing. If not otherwise obtained clinically, echocardiography will be obtained within 48 hours of admission. After a period of medical management for acutely decompensated heart failure, subjects will then have a second portable sleep apnea study (with associated pre and post-sleep blood draws) on the evening prior to discharge (approximately hospital day 5 or 6). Later, clinical outcomes such as incidence of renal dysfunction, hospital length of stay etc. will be collected from the electronic medical record. Blood samples will be processed, stored, and subsequently analyzed for high-sensitivity cardiac troponin T and I.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-80 years admitted to University of California San Diego La Jolla campus (Sulpizio Cardiovascular Center, Jacobs Medical Center, and Thornton Hospital) with acute decompensated heart failure will be identified in the emergency department, or upon admission to the cardiology or inpatient general medical services.

Exclusion Criteria:

* Known diagnosis of sleep disordered breathing and on treatment while hospitalized.
* Suspected acute coronary syndrome as determined by the primary clinical team.
* Intensive care unit level care.
* Requiring advanced heart failure therapy such as inotrope infusion, mechanical circulatory support etc.
* Intolerance of study procedures.
* Clinical attending physician refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to University of California San Diego Sulpizio Cardiovascular Center, Jacobs Medical Center, and Thornton Hospital with acutely decompensated heart failure will be identified in the emergency department, or upon admission to the cardiology or hospitalist (general medical) service.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Overnight Troponin Change Admission | 10 hours
  Overnight change in serum troponin concentration PRE vs POST sleep
Overnight Troponin Change Discharge | 10 hours
  Overnight change in serum troponin concentration PRE vs POST sleep

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Altman Clinical and Translational Research Institute, San Diego, California
  - University of California San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No